CLINICAL TRIAL: NCT07311915
Title: Propranolol Combined With Novel Endocrine Therapy and Androgen Deprivation Therapy (ADT) for Neoadjuvant Treatment in High-Risk Prostate Cancer Patients: A Multicenter, Single-Arm Clinical Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, baotai Liang, doctor, Zhongda Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZDSYLL131-P01
Record Dates: First submitted 2025-09-30; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propranolol combined with novel endocrine therapy and androgen deprivation therapy (Experimental)
  Interventions: Drug: Propranolol combined with novel endocrine therapy and androgen deprivation therapy

INTERVENTIONS:
Drug: Propranolol combined with novel endocrine therapy and androgen deprivation therapy — Patients in the group received daily oral propranolol therapy: the initial oral dose was 10 mg three times daily, with adjustments made by the clinician based on the patient's blood pressure status; concurrently administered were continuous novel endocrine therapy and androgen deprivation therapy.

SUMMARY:
Propranolol, a non-selective adrenergic beta-receptor blocker, is conventionally used to treat arrhythmias. However, recent studies have demonstrated its therapeutic efficacy in breast cancer, prostate cancer, neonatal hemangioma, and neonatal facial rhabdomyoma. Given the significant potential of neoadjuvant therapy in prostate cancer, we designed a multicenter, single-arm clinical study. This trial evaluates neoadjuvant propranolol combined with novel endocrine therapy and androgen deprivation therapy (ADT) in high-risk prostate cancer patients prior to radical prostatectomy, aiming to achieve superior curative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 85 years;

  * High-risk prostate cancer patients. High-risk prostate cancer is defined as: organ-confined high-risk/very high-risk prostate cancer and locally advanced prostate cancer. High-risk/very high-risk is specifically defined as PSA > 20 ng/mL, biopsy Gleason score ≥ 8, or clinical T stage cT2c or higher, meeting at least one of these three criteria, and without distant metastasis. Local progression typically refers to pelvic lymph node metastasis only; ③ Patients diagnosed with mild to moderate primary hypertension according to the Chinese Hypertension Prevention and Treatment Guidelines (2024 Revised Edition). Hypertension is defined as:

    * Office blood pressure ≥140/90 mmHg without antihypertensive medication; or home blood pressure ≥135/85 mmHg; or 24-hour ambulatory blood pressure ≥130/80 mmHg, with daytime blood pressure ≥135/85 mmHg and nighttime blood pressure ≥120/70 mmHg. Specifically: - Systolic blood pressure 140-159 mmHg and/or diastolic blood pressure 90-99 mmHg constitutes mild hypertension; - Systolic blood pressure 160-179 mmHg and/or diastolic blood pressure 100-109 mmHg constitutes moderate hypertension.

      * For patient screening, office blood pressure must meet any one of the following criteria:

        1. Primary hypertension patients who have not used any antihypertensive medication for at least 4 weeks prior to screening, with an average seated office blood pressure (mean of 3 measurements) of 150 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg;
        2. Patients with primary hypertension who have been on stable doses of 1-2 antihypertensive agents (including monotherapy, dual therapy, or fixed-dose combinations) for at least 4 weeks prior to screening, and who are deemed clinically suitable for switching to propranolol or nifedipine, with an average seated office blood pressure of 140 mmHg ≤ SBP < 180 mmHg and DBP < 110 mmHg; ⑤ ECOG (Eastern Cooperative Oncology Group) performance status of 0-1;

           ⑥ All patients voluntarily sign informed consent and are able to adhere to treatment and follow-up;

           ⑦ Prostate cancer biopsy specimens and surgically resected tissue are available for subsequent analysis, with sufficient tumor cell content in the pathological specimens;

           Exclusion Criteria:
* Any prior or ongoing PCa treatment, including radiotherapy, chemotherapy, ADT, etc.;

  * Individuals contraindicated for propranolol. Specifically including: 1) Patients with asthma and allergic rhinitis; 2) Patients with cardiovascular disease: sinus bradycardia, severe atrioventricular block, cardiogenic shock; 3) Patients with cardiac insufficiency; 4) Patients with hepatic impairment; 5) Patients with hypothyroidism; ③ Patients who have recently (within 3 months) taken beta-blocker medications (e.g., carvedilol, metoprolol);

    * Patients with known allergies to any medication used; ⑤ Patients on long-term antiarrhythmic drugs (e.g., amiodarone, sotalol, digoxin, verapamil, flecainide); ⑥ Patients deemed unsuitable for this clinical study by the investigator's judgment;

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | From enrollment to the end of treatment at 12 weeks
  pCR (pathological complete response) is defined as the absence of morphologically recognizable cancer in the prostate resection specimen.
Minimal Residual Disease | From enrollment to the end of treatment at 12 weeks
  MRD (Minimal Residual Disease) is defined as residual tumors with a maximum cross-sectional dimension ≤5 mm and a residual cancer burden (RCB) ≤0.25 cm³ (tumor volume ≤0.5 cm³ × tumor cell content ≤50%). Tumor volume is calculated via three-dimensional volume estimation based on the maximum cross-sectional dimension and number of cross-sections involved, with correction for tumor cell architecture.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: Yes